CLINICAL TRIAL: NCT01513928
Title: A Phase 1, Cross-Over, Single-Dose, Open-Label Study To Estimate The Relative Bioavailability Of Three Different Formulations Of PF-04937319 In Overweight And Obese Otherwise Healthy Subjects
Brief Title: A Study To Compare The Pharmacokinetics Of Different Formulations Of PF-04937319 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B1621005
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: pharmacokinetics; relative bioavailability; formulation comparison
MeSH Terms: interventions — N,N-dimethyl-5-((2-methyl-6-((5-methylpyrazin-2-yl)carbamoyl)benzofuran-4-yl)oxy)pyrimidine-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pf-04937319 — Formulation A) Pf-04937319 50 mg - administered as tablet
Drug: Pf-04937319 — Formulation B) Pf-04937319 50 mg - administered as capsule
Drug: Pf-04937319 — Formulation C) Pf-04937319 50 mg - administered as capsule

SUMMARY:
This study is designed to compare the pharmacokinetics of three different formulations of Pf-04937319

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests.
* Subjects of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 28-days after the last dose of treatment.
* Body Mass Index (BMI) of 23 to 33 kg/m2 and a total body weight >=50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (excluding untreated seasonal allergies).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Pf-04937319: Maximum plasma concentration (Cmax) | 0 - 96 hours post dose
Pf-04937319: Time for Cmax (Tmax) | 0 - 96 hours post dose
Pf-04937319: Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (AUClast) | 0 - 96 hours post dose
Pf-04937319: Area under the plasma concentration-time profile from time zero extrapolated to infinite time (AUCinf) | 0 - 96 hours post dose
Pf-04937319: terminal half-life (T1/2) | 0 - 96 hours post dose
PF-06455349: Maximum Observed Plasma Concentration (Cmax) | 0 - 96 hours post dose
PF-06455349: Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0 - 96 hours post dose
PF-06455349: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0 - 96 hours post dose
PF-06455349: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | 0 - 96 hours post dose
PF-06455349: Plasma Decay Half-Life (t1/2) | 0 - 96 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1621005&StudyName=Astudy%20To%20Compare%20The%20Pharmacokinetics%20Of%20Different%20Formulations%20Of%20PF-04937319%20In%20Healthy%20Subjects